CLINICAL TRIAL: NCT03699670
Title: eFast Diagnosis Performance in Guiding First Aid Resuscitation at the Admission of Severe Trauma Injuries
Brief Title: eFast Diagnosis Performance in Guiding First Aid Resuscitation
Acronym: eFAST Decision
Status: Completed | Type: Observational
Sponsor: University Hospital, Grenoble (Other)
Collaborators: Société Française d'Anesthésie et de Réanimation (Other)
Responsible Party: Sponsor
Other Study IDs: 38RC18.071; 2018-A00835-50 (Other: ID RCB)
Record Dates: First submitted 2018-07-06; First posted 2018-10-09 (Actual); Last update posted 2022-02-08 (Actual); Status verified 2022-02

CONDITIONS: eFast Diagnosis Performance in Guiding First Aid Resuscitation and Hemostasis
Keywords: Resuscitation; Wounds and Injuries; Ultrasonography; Radiography; Diagnostic Imaging
MeSH Terms: conditions — Wounds and Injuries

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
A lesion work-up associating clinical examination, extended focused ultrasound (eFAST including abdominal ultrasound [right upper, left upper, and suprapubic quadrant], bilateral anterior and lateral pleuropulmonary ultrasound, sub-xyphoid pericardial ultrasound, transcranial Doppler), and possibly chest and pelvis x-ray, can early diagnose the most severe traumatic lesions and guide first aid resuscitation and haemostasis. The protocol does not modify the diagnostic and therapeutic strategies applied in the participant centers.

The objective of the study is to evaluate the diagnosis performance of an initial lesion assessment by extended focused ultrasound (eFAST) (possibly associated with chest and pelvis x-ray) at the early phase of a severe trauma patient care in guiding first aid resuscitation and haemostasis.

The relevance will be judged on the therapeutic decisions taken (thoracic or pericardial drainage, thoracotomy or laparotomy, pelvic embolization, posture of a pelvic girdle, and early optimization of cerebral perfusion pressure) based on the initial ultrasound scan.

DETAILED DESCRIPTION:
Some of the severe traumatized patients who arrive alive in the hospital, are in serious hemodynamic and / or respiratory instability and need resuscitation and / or hemostasis immediate act before a complete exhaustive work-up can be realized. Usually this is a whole body CT scan. These gestures are guided by imaging examinations (extensive focused ultrasound [eFAST] +/- chest X-ray +/- pelvis X-ray) which are less accurate but faster at the patient's bedside. The ability of extended focused ultrasound to properly guide immediate resuscitation and hemostasis should be evaluated to assess effectiveness and safety of the method.

This trial is a national prospective cohort (6 French centers). Each participant will benefit from an initial lesion work-up by clinical examination, followed by an extended focused ultrasound (eFAST including abdominal ultrasound [right upper, left upper, and suprapubic quadrant], bilateral anterior and lateral pleuropulmonary ultrasound, sub-xyphoid pericardial ultrasound, transcranial Doppler), and possibly chest and pelvis frontal x-ray.

Based on clinical, radiographic and ultrasound data, the investigator will decide to perform immediate resuscitation and haemostasis gestures, or therapeutic abstention, before the realization of the complete lesion work-up by whole body CT scan.

This study could validate and strengthen the place of ultrasound in the initial severe traumatic patients' care and seems to be the continuity of the Peytel et al. research, studying new modalities of the eFAST. Our study could extend the scope and the conclusions of the Peytel et al. study to what is routinely done in the French and European Trauma Centers.

ELIGIBILITY:
Inclusion Criteria:

* Serious trauma (Grade A or B according to the TRENAU classification)
* In the emergency room of an investigator center

Exclusion Criteria:

* Patient died on site or on arrival at the emergency room
* Patient with penetrating trauma
* Patient admitted to another center and then transferred to an investigator center
* Patient referred to in Articles L1121-5 to L1121-8 of the French Code of Public Health (pregnant, parturient, breastfeeding woman, person deprived of liberty, person under legal protection).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All severe traumatized patients taken care in the emergency block of one of the investigator centers.
Sampling Method: Probability Sample
Enrollment: 510 (Actual)
Dates: Start 2018-07-03 (Actual); Primary Completion 2019-12-13 (Actual); Study Completion 2020-01-21 (Actual)

PRIMARY OUTCOMES:
Evaluation of the diagnosis performance of an initial lesion assessment by extended focused ultrasound (eFAST) at the early phase of a severe trauma patient care in guiding first aid resuscitation and haemostasis. | Through study completion, an average of 1 year
  Retrospective assessment (on whole-body CT scans data and clinical data), by a panel of experts on the legitimacy of urgent therapeutic decisions taken, following the initial injury evaluation (among a pre-selection of decisions). Assessment of presence of pericardic, intra-abdominal or pleural effusion and presence of pubic symphisis. Assessment of physiological parameters of transcranial Doppler.

SECONDARY OUTCOMES:
Evaluation of the duration of the initial lesion assessment by extended focused ultrasound (eFAST). | A Day 0
  Time measured between the arrival of the patient in the emergency room and the realization of immediate gestures of resuscitation and haemostasis
Analysis of the main outcome measure in separate criterion: US (+/- Rx). | Through study completion, an average of 1 year
  Analysis of the relevance of ultrasound vs X-rays by assessing the concordance rate between urgent therapeutic decisions and expert evaluations for each of the therapeutic modalities, taken separately
Comparison of observed mortality and predicted mortality assessed by ISS score | during patient's care, at Hour 24 and at Day 8
  Prognostic score ISS
Comparison of observed mortality and predicted mortality assessed by TRISS | during patient's care, at Hour 24 and at Day 8
  Prognostic score TRISS
Comparison of observed mortality and predicted mortality assessed by mortality evaluation | during patient's care, at Hour 24 and at Day 8
  Mortality evaluation

CONTACTS AND LOCATIONS:
Overall Officials: Pierre BOUZAT, Principal Investigator — University Hospital of Grenoble Alpes
Locations (1):
- University Hospital of Grenoble Alpes, Grenoble, Cs10217, France

REFERENCES:
- [Background] Peytel E, Menegaux F, Cluzel P, Langeron O, Coriat P, Riou B. Initial imaging assessment of severe blunt trauma. Intensive Care Med. 2001 Nov;27(11):1756-61. doi: 10.1007/s00134-001-1119-z. Epub 2001 Oct 17. PMID 11810119
- [Background] Moore CL, Copel JA. Point-of-care ultrasonography. N Engl J Med. 2011 Feb 24;364(8):749-57. doi: 10.1056/NEJMra0909487. No abstract available. PMID 21345104
- [Background] Brooks A, Davies B, Smethhurst M, Connolly J. Emergency ultrasound in the acute assessment of haemothorax. Emerg Med J. 2004 Jan;21(1):44-6. doi: 10.1136/emj.2003.005438. PMID 14734374
- [Background] Kirkpatrick AW, Sirois M, Laupland KB, Liu D, Rowan K, Ball CG, Hameed SM, Brown R, Simons R, Dulchavsky SA, Hamiilton DR, Nicolaou S. Hand-held thoracic sonography for detecting post-traumatic pneumothoraces: the Extended Focused Assessment with Sonography for Trauma (EFAST). J Trauma. 2004 Aug;57(2):288-95. doi: 10.1097/01.ta.0000133565.88871.e4. PMID 15345974
- [Background] Geeraerts T, Velly L, Abdennour L, Asehnoune K, Audibert G, Bouzat P, Bruder N, Carrillon R, Cottenceau V, Cotton F, Courtil-Teyssedre S, Dahyot-Fizelier C, Dailler F, David JS, Engrand N, Fletcher D, Francony G, Gergele L, Ichai C, Javouhey E, Leblanc PE, Lieutaud T, Meyer P, Mirek S, Orliaguet G, Proust F, Quintard H, Ract C, Srairi M, Tazarourte K, Vigue B, Payen JF; French Society of Anaesthesia; Intensive Care Medicine; in partnership with Association de neuro-anesthesie-reanimation de langue francaise (Anarlf); French Society of Emergency Medicine (Societe Francaise de Medecine d'urgence (SFMU); Societe francaise de neurochirurgie (SFN); Groupe francophone de reanimation et d'urgences pediatriques (GFRUP); Association des anesthesistes-reanimateurs pediatriques d'expression francaise (Adarpef). Management of severe traumatic brain injury (first 24hours). Anaesth Crit Care Pain Med. 2018 Apr;37(2):171-186. doi: 10.1016/j.accpm.2017.12.001. Epub 2017 Dec 27. PMID 29288841
- [Background] Jaffres P, Brun J, Declety P, Bosson JL, Fauvage B, Schleiermacher A, Kaddour A, Anglade D, Jacquot C, Payen JF. Transcranial Doppler to detect on admission patients at risk for neurological deterioration following mild and moderate brain trauma. Intensive Care Med. 2005 Jun;31(6):785-90. doi: 10.1007/s00134-005-2630-4. Epub 2005 Apr 16. PMID 15834704
- [Background] Ract C, Le Moigno S, Bruder N, Vigue B. Transcranial Doppler ultrasound goal-directed therapy for the early management of severe traumatic brain injury. Intensive Care Med. 2007 Apr;33(4):645-51. doi: 10.1007/s00134-007-0558-6. Epub 2007 Feb 27. PMID 17325830
- [Background] Shaukat NM, Copeli N, Desai P. The Focused Assessment With Sonography For Trauma (FAST) Examination And Pelvic Trauma: Indications And Limitations. Emerg Med Pract. 2016 Mar;18(3):1-20, 24; quiz 20-1. Epub 2016 Mar 1. PMID 26881977
- [Background] Bauman M, Marinaro J, Tawil I, Crandall C, Rosenbaum L, Paul I. Ultrasonographic determination of pubic symphyseal widening in trauma: the FAST-PS study. J Emerg Med. 2011 May;40(5):528-33. doi: 10.1016/j.jemermed.2009.08.041. Epub 2009 Nov 17. PMID 19926435
- [Background] Ma OJ, Mateer JR, Ogata M, Kefer MP, Wittmann D, Aprahamian C. Prospective analysis of a rapid trauma ultrasound examination performed by emergency physicians. J Trauma. 1995 Jun;38(6):879-85. doi: 10.1097/00005373-199506000-00009. PMID 7602628
- [Background] Boulanger BR, McLellan BA, Brenneman FD, Ochoa J, Kirkpatrick AW. Prospective evidence of the superiority of a sonography-based algorithm in the assessment of blunt abdominal injury. J Trauma. 1999 Oct;47(4):632-7. doi: 10.1097/00005373-199910000-00005. PMID 10528595
- See also: Related Info — http://www.cepidc.inserm.fr/